CLINICAL TRIAL: NCT03592719
Title: Motivational Interviewing to Increase PrEP Uptake (MI-PrEP)
Acronym: MI-PrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sannisha K Dale, Assistant Professor of Psychology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180516
Record Dates: First submitted 2018-07-09; First posted 2018-07-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Risk Factor
Keywords: HIV Prevention; PrEP; Black; African American; Women; Motivational Interviewing; At risk for HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-PrEP (Experimental): Participants in this arm will receive the manualized two-session intervention entitled "Motivational Interviewing to Increase PrEP Uptake"
  Interventions: Behavioral: Experimental Intervention (MI-PrEP)
- Enhanced Treatment as Usual (E-TAU) (Active Comparator): Participants in this arm will receive two sessions which entail psychoeducation on PrEP.
  Interventions: Behavioral: Enhanced Treatment as Usual (E-TAU)

INTERVENTIONS:
Behavioral: Experimental Intervention (MI-PrEP) — The experimental intervention will consist of two sessions. The first session will involve psycho-education on PrEP and Motivational Interviewing to explore ambivalence about PrEP uptake. The second session will involve Motivational Interviewing and case management to explore barriers to accessing PrEP.
  Other Names: Motivational Interviewing to Increase PrEP Uptake (MI-PrEP)
  Arms: MI-PrEP
Behavioral: Enhanced Treatment as Usual (E-TAU) — Participants assigned to the control condition will receive two sessions, both of which involve psychoeducation on PrEP.
  Arms: Enhanced Treatment as Usual (E-TAU)

SUMMARY:
The purpose of this study is to test a counseling program for Black women at high risk for HIV

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* Identify as Black and/or African American
* Age 18 or older
* Cis-gender Female
* English speaking
* Is capable of completing and fully understanding the informed consent process and the study procedures and
* Meets the Center for Disease Control's indications for PrEP use (17): (a) any sex with opposite sex partners in the past 6 months and (b) not in a monogamous partnership with a recently tested HIV-negative partner or (c) any injection of drugs not prescribed by a clinician in the past 6 months AND (d) at least one of the following: (i) infrequently uses condoms in sex with one/more partners of unknown HIV status (ii) in a sexual relationship with an HIV-positive partner or (iii) any sharing of injection/drug preparation equipment in past 6 months.

Exclusion Criteria:

* Not capable of completing/fully understanding the consent process and the study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Change in Motivation for PrEP | Baseline, Up to 6 weeks
  Motivation to use PrEP will be measured with the Contemplation Ladder and the Readiness Ruler, which assess intention to use PrEP and the perceived importance of using PrEP. The Contemplation Ladder and the Readiness Ruler each have a total score range from 0 to 10. Higher scores on the Contemplation Ladder indicate higher levels of contemplation or consideration about PrEP use. Higher scores on the Readiness Ruler indicate higher perceived importance of starting PrEP.
Change in PrEP uptake | Baseline, Up to 6 weeks
  PrEP uptake will be verified by the participants' providers.

SECONDARY OUTCOMES:
Change in Knowledge of PrEP | Baseline, Up to 6 weeks
  Knowledge of PrEP will be measured using a PrEP fact sheet, with basic information about PrEP. The PrEP Fact Sheet has a total score range of 0 to 12, with higher scores indicating higher levels of PrEP knowledge.
Change in Barriers for PrEP | Baseline, Up to 6 weeks
  Perceived barriers to PrEP uptake/usage will be measured by an adapted version of the Barriers to Care Scale, in which participants are asked about factors that make it difficult to receive PrEP related services. The Barriers to Care scale has a total score range of 7 to 28, with higher scores indicating increased difficulty regarding barriers to PrEP uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Sannisha K Dale, PhD, EdM, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No